CLINICAL TRIAL: NCT05018234
Title: Safety Monitoring for a Novel 3D Printed Mandibular Advancement Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Aaron Glick, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HSC-DB-21-0472
Record Dates: First submitted 2021-08-18; First posted 2021-08-24 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: oral appliance; sleep apnea; hypoxia
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: Noval Oral Appliance

INTERVENTIONS:
Device: Noval Oral Appliance — A scan of the mouth will be performed to make the oral device. The device will be 3D printed with Asiga UV Max printer using FDA 510(k) cleared VeriSplint OS Resin.Subjects will be will be asked to wear the oral device at night for 3 nights and fill out a survey reviewing their experience wearing the device.

SUMMARY:
The purpose of this study is to evaluate the safety profile of the novel oral appliance (OA )device and to assess patient comfort of the novel OA device.

ELIGIBILITY:
Inclusion Criteria:

* No history of obstructive sleep apnea
* No active jaw joint pain
* No active moderate to severe periodontal disease
* Presence of 12 teeth per arch

Exclusion Criteria:

* presence of severe bruxism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
safety of device as measured by the number of patients with adverse events | During the time the OA device is worn, that is, from the time of appointment 2(1 month after enrollment) to the time of appointment 3 (1 week after appointment 2)"

SECONDARY OUTCOMES:
Comfort of the novel OA device as measured by the delivery (pre care) patient feedback survey | 1 month after enrollment(appointment 2)
  Comfort will be assessed through a numerical rating scale and short answer survey that will assess comfort and user feedback while wearing the novel OA device. There are 4 questions in the survey, the first one has 5 answer choices about how the appliance fits to the teeth and ranges from very tight fit to very loose fit .The rest of the questions are rated form 1-10,a higher number indicating more comfort
Comfort of the novel OA device as measured by the post care patient feedback survey | 1 week after appointment 2(appointment 3)
  Comfort will be assessed through a numerical rating scale and short answer survey that will assess comfort and user feedback while wearing the novel OA device.There are 12 questions in the survey, the first one has 5 answer choices about how the appliance fits to the teeth and ranges from very tight fit to very loose fit .The next 8 questions are rated form 1-10,a higher number indicating more comfort, the 9th question indicates any adverse events and the last 3 questions are short answer questions describing the patient's experience with the device.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Glick, DDS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No